CLINICAL TRIAL: NCT04425031
Title: Handling Oxygenation Targets in COVID-19 Patients With Acute Hypoxaemic Respiratory Failure in the Intensive Care Unit: A Randomised Clinical Trial of a Lower Versus a Higher Oxygenation Target
Brief Title: Handling Oxygenation Targets in COVID-19
Acronym: HOT-COVID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Responsible Party: Principal Investigator, Bodil Steen Rasmussen, Clinical Professor, MD, PhD, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAUH-ICU-03; 2017-000632-34 (EudraCT Number)
Record Dates: First submitted 2020-06-05; First posted 2020-06-11 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Hypoxemic Respiratory Failure; Oxygen Toxicity
Keywords: Oxygenation; Acute Respiratory Distress Syndrome; Mechanical ventilation; Critical illness; Critical care
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Distress Syndrome; Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low oxygenation target (Experimental): Partial pressure of oxygen in arterial blood (PaO2) 8 kPa (60 mmHg)
  Interventions: Drug: Low oxygenation target
- High oxygenation target (Active Comparator): Partial pressure of oxygen in arterial blood (PaO2) 12 kPa (90 mmHg)
  Interventions: Drug: High oxygenation target

INTERVENTIONS:
Drug: Low oxygenation target — Oxygen administration to achieve a PaO2 of 8 kPa (60 mmHg) from ICU admission to ICU discharge
  Other Names: Inspired oxygen
  Arms: Low oxygenation target
Drug: High oxygenation target — Oxygen administration to achieve a PaO2 of 12 kPa (90 mmHg) from ICU admission to ICU discharge
  Other Names: Inspired oxygen
  Arms: High oxygenation target

SUMMARY:
Patients with COVID-19 and hypoxaemic respiratory failure and admitted to the intensive care unit (ICU) are treated with supplementary oxygen as a standard. However, quality of quantity evidence regarding this practise is low. The aim of the HOT-COVID trial is to evaluate the benefits and harms of two targets of partial pressure of oxygen in arterial blood (PaO2) in guiding the oxygen therapy in acutely ill adult COVID-19 patients with hypoxaemic respiratory failure at ICU admission.

DETAILED DESCRIPTION:
Acutely ill adult COVID-19 patients with hypoxaemic respiratory failure admitted to the intensive care unit (ICU) are at risk of life-threatening hypoxia, and are provided supplementary oxygen. Liberal use of supplementary oxygen may increase the number of serious adverse events including death. However, the use of supplementary oxygen therapy, and the optimal oxygenation target in COVID-19 patients have not yet been studied.

The World Health Organisation (WHO) recommends an oxygen therapy during resuscitation of COVID-19 patients to achieve an SpO2 of 94% or more, and 90% or more when stable (non-pregnant patients). The Surviving Sepsis Campaing (SSC) recommends a conservative oxygenation strategy for COVID-19 patients targeting an SpO2 no higher than 96%. Both are based on a systematic review and metanalysis from 2018, investigating the association with mortality and higher versus lower oxygenation strategies in critically ill patients in general.

COVID-19 patients admitted to the ICU and treated with positive pressure ventilation fulfil the 2012 Berlin criteria for acute respiratory distress syndrome (ARDS). Current practice regarding supplementary oxygen therapy in patients with ARDS follows the regimen used in an randomised clinical trial (RCT) from 2000 comparing lower versus higher tidal volumes; i.e. a partial pressure of arterial oxygen (PaO2) of 55-80 mmHg (7.3-10.7 kPa) or a peripheral oxygen saturation (SpO2) of 88-95%.

Of note, a recent published RCT demonstrated a lowered all-cause mortality when targeting a higher oxygenation target (PaO2: 12-14 kPa [90-105 mmHg]) compared to a lower oxygenation target (PaO2: 7.3-9.3 [55-70 mmHg]) in ARDS patients.

The quality and quantity of the current body of evidence regarding oxygenation targets in ARDS is still low.

The aim of the HOT-COVID trial is to evaluate the benefits and harms of two targets of partial pressure of oxygen in arterial blood (PaO2) in guiding the oxygen therapy in acutely ill adults COVID-19 patients with hypoxaemic respiratory failure at ICU admission.

The HOT-COVID trial is an amendment to the HOT-ICU trial (NCT03174002)

ELIGIBILITY:
Inclusion Criteria:

* Acutely admitted to the ICU AND
* Aged ≥ 18 years AND
* Receives supplemental oxygen with a flow of at least 10 L per minutes in an open system including high-flow systems OR recieves supplemental oxygen in a closed system including invasive or non-invasive ventilation or continuous positive airway pressure (CPAP)-systems AND
* Expected to receive supplemental oxygen for at least 24 hours in the ICU AND
* Having an arterial line for PaO2 monitoring AND
* Confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection (COVID-19) in the time leading to or during current hospital admission

Exclusion Criteria:

* Cannot be randomised within twelve hours after present ICU admission
* Chronic mechanical ventilation for any reason
* Use of home oxygen
* Previous treatment with bleomycin
* Organ transplant during current hospital admission
* Withdrawal from active therapy or brain death deemed imminent
* Fertile woman (< 50 years of age) with positive urine human gonadotropin (hCG) or plasma-hCG
* Carbon monoxide poisoning
* Cyanide poisoning
* Methaemoglobinaemia
* Paraquat poisoning
* Any condition expected to involve the use of hyperbaric oxygen (HBO)
* Sickle cell disease
* Consent not obtainable according to national regulations
* Previously randomised into the HOT-COVID trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 726 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
Days alive without organ support | Within 90 days
  Days alive and free from mechanical ventilation, circulatory support and renal replacement therapy

SECONDARY OUTCOMES:
90-days mortality | 90 days
  All-cause mortality 90 days after randomisation
Days alive out of the hospital | Within 90 days
  Days alive out of the hospital
Number of patients with one or more serious adverse events | Until ICU discharge, maximum 90 days
  Serious adverse events are defined as new episode of shock and new episodes of ischaemic events including myocardial or intestinal ischaemia or ischaemic stroke
1-year mortality | 1 year
  All-cause mortality 1 year after randomisation
Quality of life assessement using the EuroQoL EQ-5D-5L telephone interview | 1 year
  EQ-5D-5L 1-year after randomisation
Cognitive function 1-year after randomisation as assessed using the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) score in selected sites | 1 year
  RBANS score 1 year after randomisation at selected sites. The overall RBANS global cognition score, as well as each cognitive domain score, range from 40 to 160 with 100 ± 15 being the age-adjusted mean ± standard deviation. Higher scores indicate better performance.
Carbon monoxide diffusion capacity | 1 year
  Carbon monoxide diffusion capacity (DLCO) 1 year after randomisation at selected sites.
A health economic analysis | 90 days
  Cost-effectiveness versus cost-minimisation analyses after completion of the trial, based on the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Bodil Steen Rasmussen, MD, PhD, Principal Investigator — Aalborg University Hospital, Denmark; Bodil Steen Rasmussen, MD, PhD, Study Chair — Aalborg University Hospital, Denmark
Locations (10):
- Denmark (8):
  - Dept. of Intensive Care, Aalborg University Hospital, Aalborg
  - Dept. of Intensive Care 4131, Copenhagen University Hospital Rigshospitalet, Copenhagen
  - Dept. of Intensive Care, Herlev Hospital, Herlev
  - Dept. of Intensive Care, Hillerød Hospital, Hillerød
  - Dept. of Intensive Care, Kolding Hospital, Kolding
  - Dept. of Intensive Care, Køge Hospital, Køge
  - Randers Hospital, Randers
  - Dept. of Intensive Care, Slagelse Hospital, Slagelse
- Oslo University Hospital, Oslo, Norway
- Universitätsspital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All original records (incl. consent forms, electronic clinical report forms (eCRFs), and relevant correspondences) will be archived at trial sites for 15 years. The clean electronic trial database file will be delivered to the EudraCT Database and Zenodo data repository (https://zenodo.org/) and maintained for 15 years and anonymised if requested by the authorities.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available from June 2024 and for 10 years ahead.
Access Criteria: Access Criteria:
  Managed by the Steering Committee of the HOT-COVID trial.
URL: http://cric.nu/hot-covid

REFERENCES:
- [Background] Schjorring OL, Perner A, Wetterslev J, Lange T, Keus F, Laake JH, Okkonen M, Siegemund M, Morgan M, Thormar KM, Rasmussen BS; HOT-ICU Investigators. Handling Oxygenation Targets in the Intensive Care Unit (HOT-ICU)-Protocol for a randomised clinical trial comparing a lower vs a higher oxygenation target in adults with acute hypoxaemic respiratory failure. Acta Anaesthesiol Scand. 2019 Aug;63(7):956-965. doi: 10.1111/aas.13356. Epub 2019 Mar 18. PMID 30883686
- [Background] Barbateskovic M, Schjorring OL, Jakobsen JC, Meyhoff CS, Rasmussen BS, Perner A, Wetterslev J. Oxygen supplementation for critically ill patients-A protocol for a systematic review. Acta Anaesthesiol Scand. 2018 Aug;62(7):1020-1030. doi: 10.1111/aas.13127. Epub 2018 Apr 30. PMID 29708586
- [Background] Barbateskovic M, Schjorring OL, Russo Krauss S, Jakobsen JC, Meyhoff CS, Dahl RM, Rasmussen BS, Perner A, Wetterslev J. Higher versus lower fraction of inspired oxygen or targets of arterial oxygenation for adults admitted to the intensive care unit. Cochrane Database Syst Rev. 2019 Nov 27;2019(11):CD012631. doi: 10.1002/14651858.CD012631.pub2. PMID 31773728
- [Background] Rasmussen BS, Perner A, Wetterslev J, Meyhoff CS, Schjorring OL. Oxygenation targets in acutely ill patients: still a matter of debate. Lancet. 2018 Dec 8;392(10163):2436-2437. doi: 10.1016/S0140-6736(18)32201-3. No abstract available. PMID 30527413
- [Background] Schjorring OL, Klitgaard TL, Perner A, Wetterslev J, Lange T, Keus F, Laake JH, Morgan M, Backlund M, Siegemund M, Thormar KM, Rasmussen BS. The handling oxygenation targets in the intensive care unit (HOT-ICU) trial: Detailed statistical analysis plan. Acta Anaesthesiol Scand. 2020 Jul;64(6):847-856. doi: 10.1111/aas.13569. Epub 2020 Mar 4. PMID 32068884
- [Result] Nielsen FM, Klitgaard TL, Bruun NH, Moller MH, Schjorring OL, Rasmussen BS. Lower or higher oxygenation targets in the intensive care unit: an individual patient data meta-analysis. Intensive Care Med. 2024 Aug;50(8):1275-1286. doi: 10.1007/s00134-024-07523-3. Epub 2024 Jul 11. PMID 38990335
- [Result] Nielsen FM, Klitgaard TL, Siegemund M, Laake JH, Thormar KM, Cole JM, Aagaard SR, Bunzel AG, Vestergaard SR, Langhoff PK, Pedersen CH, Hejlesen JO, Abdelhamid S, Dietz A, Gebhard CE, Zellweger N, Hollinger A, Poulsen LM, Weihe S, Andersen-Ranberg NC, Pedersen UG, Mathiesen O, Andreasen AS, Brix H, Thomsen JJ, Petersen CH, Bestle MH, Wichmann S, Lund MS, Mortensen KM, Brand BA, Haase N, Iversen SA, Marcussen KV, Brochner AC, Borup M, Grofte T, Hildebrandt T, Kjaer MN, Engstrom J, Lange T, Perner A, Schjorring OL, Rasmussen BS; HOT-COVID Trial Group. Lower vs Higher Oxygenation Target and Days Alive Without Life Support in COVID-19: The HOT-COVID Randomized Clinical Trial. JAMA. 2024 Apr 9;331(14):1185-1194. doi: 10.1001/jama.2024.2934. PMID 38501214
- [Derived] Nielsen FM, Klitgaard TL, Granholm A, Lange T, Perner A, Schjorring OL, Rasmussen BS. Lower or Higher Oxygenation Targets in Patients With COVID-19 in the ICU: A Secondary Bayesian Analysis of the Handling Oxygenation Targets in COVID-19 Trial. Chest. 2025 Mar;167(3):757-767. doi: 10.1016/j.chest.2024.08.055. Epub 2024 Sep 18. PMID 39303806
- See also: Link to the HOT-COVID website — http://cric.nu/hot-covid